CLINICAL TRIAL: NCT06083675
Title: Efficacy and Safety of First Line Use of Oral Semaglutide 25 mg or 50 mg Once Daily Versus Empagliflozin 25 mg or Versus Metformin 2000 mg in Newly Diagnosed Treatment naïve Patients With Type 2 Diabetes
Brief Title: Research Study to Compare Semaglutide Tablets With Empagliflozin or Metformin Tablets in People With Type 2 Diabetes
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Due to internal reprioritization, trial was cancelled.
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NN9924-7663; U1111-1291-4976 (Other: World Health Organization (WHO))
Record Dates: First submitted 2023-10-09; First posted 2023-10-16 (Actual); Last update posted 2024-02-26 (Actual); Status verified 2024-02

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — semaglutide; empagliflozin; Metformin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Semaglutide 25 mg (Experimental): Participants will receive 25 mg oral semaglutide once daily in maintenance period after dose escalation period.
  Interventions: Drug: Semaglutide
- Semaglutide 50 mg (Experimental): Participants will receive 50 mg oral semaglutide once daily in maintenance period after dose escalation period.
  Interventions: Drug: Semaglutide
- Empagliflozin 25 mg (Experimental): Participants will 25 mg empagliflozin oral once daily in maintenance period after dose escalation period.
  Interventions: Drug: Empagliflozin
- Metformin 2000 mg (Experimental): Participants will receive metformin 1000 mg orally twice daily (total 2000 mg) in maintenance period after dose escalation period.
  Interventions: Drug: Metformin

INTERVENTIONS:
Drug: Semaglutide — Administered as oral tablets.
  Arms: Semaglutide 25 mg; Semaglutide 50 mg
Drug: Empagliflozin — Administered as oral tablets.
  Arms: Empagliflozin 25 mg
Drug: Metformin — Administered as oral tablets.
  Arms: Metformin 2000 mg

SUMMARY:
This study compares the medicines semaglutide with empagliflozin or metformin in people with newly diagnosed type 2 diabetes. This study will look mainly at how well participant's blood sugar and body weight are controlled when they are taking the study medicines. Participants will either get semaglutide tablets, empagliflozin tablets or metformin tablets. Which treatment participants will get is decided by chance. Currently, doses of 3 milligram (mg), 7 mg and 14 mg semaglutide tablets (Rybelsus) can be prescribed in some countries. 25 mg and 50 mg semaglutide tablets are new doses. 10 mg and 25 mg empagliflozin tablets (Jardiance) can be prescribed in some countries. 500 mg metformin tablets (STADA) can be prescribed in some countries. Participants will get 1 to 4 tablets per day for 104 weeks. The study will last for about 2 years and 7 weeks (111 weeks). Participants should not have been treated for weight management 90 days before screening or never been treated with any medicine for type 2 diabetes (except diabetes during pregnancy) before screening. Women cannot take part if pregnant, breast-feeding or plan to get pregnant during the study period.

ELIGIBILITY:
Inclusion Criteria:

* Male or female.
* Age ≥18 and <60 years at the time of signing the informed consent.
* Diagnosed with type 2 diabetes mellitus within 24 months from the day of screening.
* HbA1c of 7.0-10.0% (53-86 millimoles per mole [mmol/mol])
* Body mass index ≥25.0 kilogram per square meter (kg/m^2)

Exclusion Criteria:

* Treatment with any medication for the indication of diabetes. Prior insulin treatment for gestational diabetes is allowed.
* Treatment with any medication for the indication of weight management 90 days prior to screening.
* Renal impairment measured as estimated glomerular filtration rate (eGFR) <60 milliliters per minute per 1.73 meter sqaure (mL/min/1.73 m^2) at screening.
* Uncontrolled and potentially unstable diabetic retinopathy or maculopathy. Verified by a fundus examination performed within 90 days before screening or in the period between screening and randomisation. Pharmacological pupil-dilation is a requirement unless using a digital fundus photography camera specified for non-dilated examination.
* C-peptide <1.5 nanograms per milliliter (ng/mL) at screening.
* Positive insulinoma associated-protein 2 (IA-2) antibodies ≥7.5 Units/mL or anti-glutamic acid decarboxylase (anti-GAD) antibodies greater than (>) 5.0 international units per milliliter (IU/mL).
* Impaired liver function, defined as Alanine aminotransferase (ALT) ≥2.5 times or Bilirubin >1.5 times upper normal limit at screening.
* History of major surgical procedures involving the stomach potentially affecting absorption of trial products (example subtotal or total gastrectomy, sleeve gastrectomy, gastric bypass surgery) or current presence of gastrointestinal implant.
* Presence of clinically significant gastrointestinal disorders affecting absorption of drugs and/or nutrients, as judged by the investigator.
* Any contraindications for empagliflozin or metformin according to local labelling at the investigator's discretion

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2024-01-26 (Estimated); Primary Completion 2025-01-24 (Estimated); Study Completion 2027-05-28 (Estimated)

PRIMARY OUTCOMES:
Change in glycated haemoglobin (HbA1c) | From randomisation (week 0) to week 52
  Measured in Percentage (%)-points.

SECONDARY OUTCOMES:
Change in body weight | From randomisation (week 0) to week 52
  Measured in kilograms (kg).
Change in fasting plasma glucose (FPG) | From randomisation (week 0) to week 52
  Measured in millimoles per liter (mmol/L).
Change in 7 point self measured plasma glucose (SMPG) mean profile | From randomisation (week 0) to week 52
  Measured in mmol/L.
Change in 7-point self-measured plasma glucose (SMPG) mean post prandial increments | From randomisation (week 0) to week 52
  Measured in mmol/L.
Relative change in body weight | From randomisation (week 0) to week 52
  Measured in Percentage (%).
Change in waist circumference | From randomisation (week 0) to week 52
  Measured in centimeters (cm).
HbA1c less than or equal to (≤) 6.5% (Yes/No) | At week 52
  Measured as count of participants.
HbA1c less than (<) 7% (Yes/No) | At week 52
  Measured as count of participants.
Body weight reduction greater than equal to ( ≥) 5% (Yes/No) | At week 52
  Measured as count of participants.
Body weight reduction ≥10% (Yes/No) | At week 52
  Measured as count of participants.
Body weight reduction ≥15% (Yes/No) | At week 52
  Measured as count of participants.
HbA1c <7.0% and body weight reduction ≥5% (Yes/No) | At week 52
  Measured as count of participants.
Change in systolic blood pressure | From randomisation (week 0) to week 52
  Measured in millimeters of mercury (mmHg).
Change in diastolic blood pressure | From randomisation (week 0) to week 52
  Measured in mmHg.
Change in High-sensitivity C-reactive protein (hsCRP) | From randomisation (week 0) to week 52
  Measured in milligrams per liter (mg/L).
Time to rescue medication | From randomisation (week 0) to week 104
  Measured in days.
Change in HbA1c | From randomisation (week 0) to week 104
  Measured in %-points.
Change in body weight | From randomisation (week 0) to week 104
  Measured in kg.
Change in FPG | From randomisation (week 0) to week 104
  Measured in mmol/L.
Change in 7 point SMPG mean profile | From randomisation (week 0) to week 104
  Measured in mmol/L.
Change in 7-point SMPG mean post prandial increments | From randomisation (week 0) to week 104
  Measured in mmol/L
Relative change in body weight | From randomisation (week 0) to week 104
  Measured in Percentage.
Change in waist circumference | From randomisation (week 0) to week 104
  Measured in cm.
HbA1c ≤6.5% (Yes/No) | At week 104
  Measured as count of participants.
HbA1c <7.0% (Yes/No) | At week 104
  Measured as count of participants.
Body weight reduction ≥5% (Yes/No) | At week 104
  Measured as count of participants.
Body weight reduction ≥10% (Yes/No) | At week 104
  Measured as count of participants.
Body weight reduction ≥15% (Yes/No) | At week 104
  Measured as count of participants.
HbA1c <7.0% and body weight reduction ≥5% (Yes/No) | At week 104
  Measured as count of participants.
Change in systolic blood pressure | From randomisation (week 0) to week 104
  Measured in mmHg.
Change in diastolic blood pressure | From randomisation (week 0) to week 104
  Measured in mmHg.
Change in hsCRP | From randomisation (week 0) to week 104
  Measured in mg/L.
Treatment emergent adverse events | From randomisation (week 0) to week 52
  Measured as count of events.
Number of severe (level 3) or clinically significant (level 2) hypoglycaemic episodes | From randomisation (week 0) to week 52
  Measured as count of episodes.
Treatment emergent adverse events | From randomisation (week 0) to follow-up visit (week 109)
  Measured as count of events.
Number of severe (level 3) or clinically significant (level 2) hypoglycaemic episodes | From randomisation (week 0) to follow-up visit (week 109)
  Measured as count of episodes.
Change in Control of Eating Questionnaire (CoEQ) score - Craving Control domain | From randomisation (week 0) to week 52
  CoEQ is a 19-item multidimensional patient reported outcome (PRO) that assesses the experience of hunger, satiety, and severity and type of food cravings. CoEQ consists of 4 subscales that measure craving control (5 items), positive mood (4 items), craving for sweet (4 items), craving for savoury food (4 items), and 2 single items that address hunger and satiety. Each item is evaluated on a 0-10 (i.e., 11-point) numeric rating scale. The total score for each subscale is calculated as the sum of the item scores divided by the number of items in the subscale. Scores ranges are thus: Craving Control 0-50/5 = 0-10); Positive Mood (0-40/4 = 0-10); Craving Sweet (0-40/4 = 0-10); Craving Savoury food (0-40/4 = 0-10); single items that address hunger and satiety (0-10). For the craving control subscale, the subscale score is reversed so that a higher score represents a greater level of craving control.
Change in CoEQ score - Craving for Savory domain | From randomisation (week 0) to week 52
  CoEQ is a 19-item multidimensional PRO that assesses the experience of hunger, satiety, and severity and type of food cravings. CoEQ consists of 4 subscales that measure craving control (5 items), positive mood (4 items), craving for sweet (4 items), craving for savoury food (4 items), and 2 single items that address hunger and satiety. Each item is evaluated on a 0-10 (i.e., 11-point) numeric rating scale. The total score for each subscale is calculated as the sum of the item scores divided by the number of items in the subscale. Scores ranges are thus: Craving Control 0-50/5 = 0-10); Positive Mood (0-40/4 = 0-10); Craving Sweet (0-40/4 = 0-10); Craving Savoury food (0-40/4 = 0-10); single items that address hunger and satiety (0-10). For the craving savoury food subscale, higher score represents a greater level of craving.
Change in Impact of Weight on Quality of Life-Lite Clinical Trials (IWQOL-Lite-CT) score - Physical function domain | From randomisation (week 0) to week 52
  IWQOL-Lite-CT measures weight-related physical and psychosocial functioning. The measure consists of 20 items yielding 3 composite scores, and 1 total score. Higher scores indicate better levels of functioning. Composite scores (score range): Physical composite (0-100), Psychosocial composite (0 100), Physical Function composite (0-100). Total score range (0-100).
Change in American Heart Association (AHA) Life's Simple 7 summary score | From randomisation (week 0) to week 52
  The AHA recommends focusing on 7 cardiovascular health factors (smoking, BMI, physical activity, diet, total cholesterol, blood pressure, and fasting blood glucose) for early or primary prevention of cardiovascular disease. The 7 health factors are each categorized as ideal, intermediate, or poor. Scales range from 0 (minimum) to 14 (maximum). Higher score represents a greater level of health.
Change in CoEQ score - Craving Control domain | From randomisation (week 0) to week 104
  CoEQ is a 19-item multidimensional PRO that assesses the experience of hunger, satiety, and severity and type of food cravings. CoEQ consists of 4 subscales that measure craving control (5 items), positive mood (4 items), craving for sweet (4 items), craving for savoury food (4 items), and 2 single items that address hunger and satiety. Each item is evaluated on a 0-10 (i.e., 11-point) numeric rating scale. The total score for each subscale is calculated as the sum of the item scores divided by the number of items in the subscale. Scores ranges are thus: Craving Control 0-50/5 = 0-10); Positive Mood (0-40/4 = 0-10); Craving Sweet (0-40/4 = 0-10); Craving Savoury food (0-40/4 = 0-10); single items that address hunger and satiety (0-10). For the craving control subscale, the subscale score is reversed so that a higher score represents a greater level of craving control.
Change in CoEQ score - Craving for Savory domain | From randomisation (week 0) to week 104
  CoEQ is a 19-item multidimensional PRO that assesses the experience of hunger, satiety, and severity and type of food cravings. CoEQ consists of 4 subscales that measure craving control (5 items), positive mood (4 items), craving for sweet (4 items), craving for savoury food (4 items), and 2 single items that address hunger and satiety. Each item is evaluated on a 0-10 (i.e., 11-point) numeric rating scale. The total score for each subscale is calculated as the sum of the item scores divided by the number of items in the subscale. Scores ranges are thus: Craving Control 0-50/5 = 0-10); Positive Mood (0-40/4 = 0-10); Craving Sweet (0-40/4 = 0-10); Craving Savoury food (0-40/4 = 0-10); single items that address hunger and satiety (0-10). For the craving savoury food subscale, higher score represents a greater level of craving.
Change in IWQOL-Lite-CT score - Physical function domain | From randomisation (week 0) to week 104
  IWQOL-Lite-CT measures weight-related physical and psychosocial functioning. The measure consists of 20 items yielding 3 composite scores, and 1 total score. Higher scores indicate better levels of functioning. Composite scores (score range): Physical composite (0-100), Psychosocial composite (0 100), Physical Function composite (0-100). Total score range (0-100).
Change in AHA Life's Simple 7 summary score | From randomisation (week 0) to week 104
  The AHA recommends focusing on 7 cardiovascular health factors (smoking, BMI, physical activity, diet, total cholesterol, blood pressure, and fasting blood glucose) for early or primary prevention of cardiovascular disease. The 7 health factors are each categorized as ideal, intermediate, or poor. Scales range from 0 (minimum) to 14 (maximum). Higher score represents a greater level of health.

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Transparency (dept. 2834), Study Director — Novo Nordisk A/S
Locations (100):
- Hillcrest Family Health Center, Waco, Texas, United States
- Brazil (4):
  - Instituto de Ciências Farmacêuticas, Goiânia, Goiás
  - Núcleo de Pesquisa Clínica do Rio Grande do Sul Ltda., Porto Alegre, Rio Grande do Sul
  - CPQuali Pesquisa Clínica Ltda, São Paulo, São Paulo
  - CPCLIN - Centro de Pesquisas Clínicas, São Paulo, São Paulo
- Bulgaria (7):
  - Individual Practice For Specialized Outpatient Medical Care Doctor Miglena Rizova Ltd., Kyustendil
  - Diagnostic-Consultative Centre "Sveti Georgi" Eood, Plovdiv
  - "Aipsomcemd - Dr. Petya Georgieva" Eood, Plovdiv
  - ''Aipsomcidemd - Dr. Lilyana Bodurova-Troharova" Eood, Samokov
  - "Medical center Medishtit Velisia" OOD, Stara Zagora
  - Diagnostic Consulting Center 1 Velingrad EOOD, Velingrad
  - MHAT- Hristo Botev AD, Vratsa
- Croatia (5):
  - Poliklinika SLAVONIJA OSIJEK, Osijek, County of Osijek-Baranja
  - Opca bolnica Karlovac, Karlovac
  - Specijalna bolnica Krapinske Toplice - Endokrinologija, Krapinske Toplice
  - Opca bolnica Pula, Pula
  - Specijalna bolnica Medico, Rijeka
- Greece (10):
  - Iatriko Psychicou Private Clinic, Athens
  - "Laiko" General Hospital of Athens, Athens
  - Iatriko Athinon (Athens Medical Canter), Athens
  - Iatriko Athinon 'Palaiou Falirou', Athens
  - University Hospital of Athens ATTIKON, Haidari-Athens
  - University General Hospital of Ioannina,Internal Medicine, Ioannina
  - General Hospital of Thessaloniki 'G. Gennimatas, Thessaloniki
  - EUROMEDICA Gen Clinic The/ki, Endocrin,Metabolism,Diabetes, Thessaloniki
  - "Thermi" Private Hosital, Thessaloniki
  - General Hospital of Thessaloniki "G.Papanikolaou", Thessaloniki
- Hungary (2):
  - ClinDiab Egészségügyi Szolgáltató és Kereskedelmi Kft., Budapest
  - Belinus Bt., Debrecen
- India (31):
  - Osmania General Hospital, Hyderabad, A.P.
  - Endolife Specialty Hospitals, Guntur, Andhra Pradesh
  - Yalamanchi Hospitals and Research centres pvt ltd, Vijaywada, Andhra Pradesh
  - Navneeth Memorial Hospital, Ahmedabad, Gujarat
  - Govt Medical College, Vadodara, Gujarat
  - Ramaiah Memorial Hospital, Bangalore, Karnataka
  - Lifecare Hospital and Research Centre, Bangalore, Karnataka
  - K R Hospital, Mysuru, Karnataka
  - TOTALL Diabetes Hormone Institute, Indore, Madhya Pradesh
  - Goa Medical College, Goa, Maharashtra
  - Excel Endocrine Centre, Kolhāpur, Maharashtra
  - Seth GS Medical College & KEM Hospital, Mumbai, Maharashtra
  - BSES MG hospital, Mumbai, Maharashtra
  - Ashirwad Hospital and Research Centre, Thane, Maharashtra
  - Acharya Vinoba Bhave Rural Hospital, Sawangi Meghe, Wardha, Wardha, Maharashtra
  - Maulana Azad Medical College, Delhi, New Delhi
  - Dayanand Medical College & Hospital_Ludhiana, Ludhiana, Punjab
  - Jawahar Lal Nehru Govt. Medical College, Ajmer, Rajasthan
  - Diabetes, Thyroid and Endocrine Centre, Jaipur, Rajasthan
  - M.V.Hospital for Diabetes Pvt. Ltd., Chennai, Tamil Nadu
  - Gandhi Hospital & Medical college, Hyderabad, Telangana
  - Yashoda hospital, Hyderabad, Telangana
  - Medanta Lucknow Hospital, Lucknow, Uttar Pradesh
  - BP Poddar Hospital, Kolkata, West Bengal
  - Swasthya Diabetes Care, Ahmedabad
  - Aligarh Muslim University, Aligarh
  - Sparsh Hospital, Bhubaneshwar, Bhubaneshwar
  - All India Institute of Medical Sciences (AIIMS), Nagpur, Maharashtra
  - JIPMER, Puducherry
  - Lifepoint Multispecialty Hospital, Pune
  - Mahatma Gandhi Memorial Hospital, Sherpura, Warangal
- Malaysia (8):
  - Hospital Miri, Sarawak, Miri
  - Klinik Kesihatan Kuang, Rawang, Selangor
  - Klinik Kesihatan Bintulu, Bintulu
  - Klinik Kesihatan Greentown Ipoh, Ipoh
  - Klinik Kesihatan Cheras Baru, Kuala Lumpur
  - Hospital Melaka, Malacca
  - Hospital Seri Manjung, Seri Manjung
  - Hospital Sultan Haji Ahmad Shah, Temerloh,Pahang
- Mexico (3):
  - Eme Red Hospitalaria, Mérida, Yucatán
  - Medical Care and Research S. A de C.V, Mérida, Yucatán
  - FAICIC S. de R.L. de C.V., Veracruz
- Poland (12):
  - ETG Siedlce, Siedlce, Masovian Voivodeship
  - NZOZ Vita-Diabetica Malgorzata Buraczyk, Bialystok, Podlaskie Voivodeship
  - Centrum Medyczne Intercor Sp. z o.o., Bydgoszcz
  - Diab Serwis Popenda Spółka Jawna, Chorzów
  - NZOZ Euromedica, Grudziądz
  - Centra Medyczne Medyceusz Sp. z o.o., Lodz
  - Etyka Ośrodek Badań Klinicznych Tomasz Pesta S.K.A., Olsztyn
  - ENDOPRACTICA W.Beker, D.Mielczarek, P.Mielczarek, J.Struzik spółka cywilna, Opole
  - NZOZ NEURO-KARD Ilkowski i Partnerzy Spółka Partnerska Lekarzy, Poznan
  - Centrum Medyczne Oporow, Wroclaw
  - Trialmed CRS, Piotrkow Trybunalski, Łódź Voivodeship
  - Clinmedica Research sp. z o.o., Skierniewice, Łódź Voivodeship
- Romania (7):
  - Institutul National De Diabet Nutritie Si Boli Metabolice Prof.Dr.N.Paulescu Bucuresti- Ion Movila, Bucharest, Bucurestii
  - Sc Mediab Srl, Târgu Mureş, Mureș County
  - Clinica Grivitei 224 S.R.L., Brăila
  - SC Nutrilife SRL, Bucharest
  - Diabet Med SRL, Bucharest
  - S.C. Dianutrilife Medica S.R.L., Ploieşti
  - Clinica Korall S.R.L. Satu Mare, Satu Mare
- Serbia (3):
  - Healthcare centre Zvezdara, Belgrade, RS
  - Healthcare centre Kragujevac, Kragujevac, RS
  - Healthcare centre Nis, Niš, RS
- Thailand (7):
  - Siriraj Hospital, Bangkok Noi, Bangkok
  - Thammasat University Hospital, Klong Luang, Changwat Pathum Thani
  - Rajavithi Hospital, Bangkok
  - Ramathibodi Hospital, Bangkok
  - Maharaj Nakorn Chiang Mai Hospital, Chiang Mai
  - Srinagarind Hospital, Khon Kaen
  - Songklanagarind Hospital, Songkhla

IPD SHARING:
Plan to Share IPD: Yes
According to the Novo Nordisk disclosure commitment on novonordisk-trials.com
URL: http://novonordisk-trials.com